CLINICAL TRIAL: NCT00615511
Title: Efficacy of Pregnenolone in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Jason Kim, Assistant Professor of Psychiatry, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRE0504007841; 05T-658 (Other Grant/Funding Number: Stanley Medical Research Institute)
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; negative symptoms; cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Approximately one third of subjects
  Interventions: Dietary Supplement: placebo pregnenolone
- Pregnenolone (Experimental)
  Interventions: Dietary Supplement: pregnenolone

INTERVENTIONS:
Dietary Supplement: placebo pregnenolone — Sugar pill, taken twice a day
  Arms: placebo
Dietary Supplement: pregnenolone — 500mg in tablet form taken orally twice a day
  Arms: Pregnenolone

SUMMARY:
Four-month trial of pregnenolone or placebo, as an additional medication, to treat negative symptoms and cognitive decline in schizophrenia. After four months the scores on the negative symptom scale should be lower and the scores on the cognitive tests should be higher than they were at study entry, compared with people who do not take any additional medication.

DETAILED DESCRIPTION:
Pregnenolone is a steroid health supplement which is readily available in health food stores. We are using it in this study at higher doses than you would normally take as a health supplement because preliminary studies have indicated that negative symptoms improve and certain aspects of cognition improve at these doses. We do not require you to stop your existing treatment in order to enter the study. After four months we will test your symptoms and cognition and ask if you would like to continue taking pregnenolone, at no cost, in a follow-up study designed to determine the long-term costs and benefits of taking pregnenolone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Diagnosis of schizophrenia or schizoaffective disorder
* No new medication for past 3 months and stable dose for past 4 weeks
* SANS (Negative symptom) score of 20 or above

Exclusion Criteria:

* Significant dementia or head trauma.
* Seizure during past year.
* Substance dependence in past 6 months or positive urine drug screen.
* History of hormone-sensitive cancer such as breast, testicular, prostate, ovarian or uterine cancers.
* Steroid metabolism disorder, e.g.Cushings or Addison's disease.
* Taking steroids other than birth control or post-menopausal hormones.
* Women who are pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
SANS - Scale for the Assessment of Negative Symptoms | every month for 4 months

SECONDARY OUTCOMES:
Quality of Life | every two months for four months

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Kim, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - University of Medicine & Dentistry of New Jersey- University Behavioral HealthCare, Piscataway, New Jersey
  - Weill Medical College of Cornell University, New York, New York
  - Weill Medical College of Cornell University, White Plains, New York